CLINICAL TRIAL: NCT00238927
Title: Multicenter Randomised Controlled Trial of Episodic Fluticasone Versus Placebo in Viral-induced Asthma in Children
Brief Title: Clinical Trial of Fluticasone Versus Placebo at the Onset of a Cold for Children With Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Medical Research Council of Canada (Other)
Responsible Party: Principal Investigator, Francine Ducharme, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FAP30006; MRC/PMAC program
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Asthma
Keywords: asthma; preschool; viral; upper respiratory track infection; fluticasone; inhaled corticosteroids; placebo; exacerbations; severity; safety; growth; bone mineral density; adrenal function; rescue beta2-agonists
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: inhaled fluticasone 750 mcg/day twice daily until 2 days without symptoms (maximum 15 consecutive days)

SUMMARY:
The purpose of this study is to determine, in children aged 1 to 6 years with recurrent asthma induced by upper respiratory tract infections (URTI), whether the administration of high doses of inhaled fluticasone started at the onset of symptoms of a cold will result in a reduced severity and shorter duration of asthma exacerbations and will not be associated with reduced growth velocity, osteopenia, and adrenal suppression.

DETAILED DESCRIPTION:
Preschool-aged children, who represent over half of asthmatics presenting to a pediatric emergency department with acute asthma, also account for most hospital admissions for pediatric asthma. More than 80% of exacerbations of preschool-aged children are triggered by upper respiratory tract infections (URTIs). Current management of this condition is clearly unsatisfactory. In most cases, there is a 24-48 hour delay between the first signs of a viral infection and the onset of asthmatic symptoms, suggesting that a window of opportunity where an intervention could be initiated to alter the severity of the asthma exacerbation. Prior trials testing chronic inhaled steroids throughout the viral season failed to demonstrate any benefit while those examining episodic inhaled steroids at onset of URTI reported a modest benefit on duration and severity of symptoms. The selection of children with mild exacerbations, the small sample size, the cross-over design, the short study period, and the relatively low doses of inhaled steroids may have limited the magnitude of observed benefits attributable to episodic treatment.

The aim of this multicentre double-blind parallel-group placebo-controlled randomized trial is to compare the effectiveness of high doses (750 ug bid) of inhaled fluticasone with HFA propellant versus placebo started at the onset of a viral illness in attenuating the severity and duration of URTI-induced asthma in young children during a 12-month study period. Children aged 1 to 6 years with at least 2 URTI-induced asthma of moderate severity, i.e. requiring a short course of systemic steroids, in the previous 12 months or 1 in the previous 6 months, and no inter-current symptoms will be selected for inclusion. Fluticasone 250 ug or placebo will be administered at a dose of 3 puffs BID from the onset of viral illness until 48 hours without asthma symptoms for a maximum of 10 days. This dose was chosen to approach the efficacy of systemic steroids with significantly less adverse effects. Inhaled salbutamol will be administered as bronchodilator on an "as needed" basis for relief of asthma symptoms at a dose of 2 to 4 puffs of 100 ug at 4-hour interval or longer. A 7-day run-in period will serve to (1) establish the absence of chronic symptoms and the infrequent use of salbutamol and (2) obtain confirmation of eligibility by the pharmacy reports of all corticosteroid preparation dispensed in the preceding 12 months. Eligible children will receive baseline measurement of IgE as measure of atopy, varicella antibodies and of the safety parameters, including height, basal cortisol, and lumbar bone density. Children will then be randomly allocated to one of the two treatments in blocks of 4 with stratification on type of spacer (with mask or with mouthpiece) and recruitment site. Children will be followed every 3±1/2 months by the site investigators or delegates until the end of the 12-month study period. The primary endpoint is the proportion of URTIs in each group requiring treatment with systemic corticosteroids as confirmed by review of medical records and pharmacy records of prescriptions dispensed. Secondary endpoints include other measures of the severity and duration of exacerbations, adjusted for the number of URTIs experienced by each child during the study period. Compliance with the study drug and the use of salbutamol (an important measure of severity) will be documented by the Doser, a device attached to the study inhalers which records, in a blinded mode, the date and number of doses administered over a 45-day period. The safety profile will be examined with the growth velocity, the basal cortisol, and the change in lumbar bone density between baseline and the end of the study period.

A clinically important reduction in the severity and duration of viral-induced asthma will lead to other trials to establish the lowest effective dose of fluticasone. If no adverse effects on growth, bone density, and adrenal function are detected with the tested dose, safety may be assumed at lower doses. An absence of benefit will lead to the abandonment of this frequently used treatment strategy to consider alternative therapies for young children with URTI-induced asthma, who contribute to a marked proportion of health care spending.

An upper respiratory tract infection is defined as rhinorrhea, nasal congestion, sore throat, ear ache, with or without fever, lasting >=48 hours.

URTI-induced asthma is defined by wheezing in association with an URTI.

ELIGIBILITY:
Inclusion Criteria:

* (1) Children aged 1-6 years,
* (2) they had at least 2 documented episodes of URTI-induced asthma requiring systemic (i.e., oral, intravenous, or intramuscular) corticosteroids in the previous 12 months or 1 episode in the previous 6 months,
* (3) no intercurrent symptoms (i.e., cough, wheezing, or observed dyspnea) documented for at least 7 days between wheezing episodes,
* (4) no suspicion of allergy to pollen or perennial allergens, and
* (5) caregivers have a good understanding of French or English

Exclusion Criteria:

* (a) other chronic diseases such as cystic fibrosis, bronchopulmonary dysplasia, cardiac disease, kidney disease, gastro-oesophageal reflux requiring treatment,
* (b) intake, in the 21 days preceding randomization, of inhaled, nasal, or oral corticosteroids, leukotriene antagonists, cromolyn, nedocromyl, or ketotifen, -(c) prior intubation for an asthma exacerbation.

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150
Dates: Start 1999-11; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The proportion of upper respiratory tract infections (URTIs) in each group requiring treatment with systemic corticosteroids as confirmed by review of medical records and pharmacy records of prescriptions dispensed.

SECONDARY OUTCOMES:
Rate of unscheduled visits for asthma to an acute care setting adjusted for the number of upper respiratory tract infections (URTIs).
Rate of hospital admissions for asthma adjusted for the number of URTIs.
Maximum and mean number of puffs of ß2-agonists/day during URTI illness.
Peak and mean symptom scores during URTI illness
The mean # of days/URTI during which rescue ß2-agonists were used for asthma symptoms.
The mean # of days/URTI during which asthma symptoms were observed
growth velocity from baseline to endpoint
change in bone mineral density between baseline and endpoint
proportion of osteopenia at endpoint
change from baseline in hypothalamo-pituitary adrenal function (basal cortisol) at endpoint
proportion of adrenal suppression at endpoint
proportion of treatment interruption due to perceived ineffectiveness in each group

CONTACTS AND LOCATIONS:
Overall Officials: Francine M. Ducharme, MD, MSc, Principal Investigator — CHUS Ste-Justine Hospital
Locations (5):
- Canada (5):
  - Hopital Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Hopital Maisonneuve-Rosemont, Montreal, Quebec
  - Centre Pédiatrique La Courte Échelle, Repentigny, Quebec
  - Centre Hospitalier Universitaire de Sherbrooke, Sherbrooke, Quebec

REFERENCES:
- [Derived] Ducharme FM, Lemire C, Noya FJ, Davis GM, Alos N, Leblond H, Savdie C, Collet JP, Khomenko L, Rivard G, Platt RW. Preemptive use of high-dose fluticasone for virus-induced wheezing in young children. N Engl J Med. 2009 Jan 22;360(4):339-53. doi: 10.1056/NEJMoa0808907. PMID 19164187